CLINICAL TRIAL: NCT04980976
Title: C-MAC Videolaryngoscope for Insertion of a Transesophageal Echocardiography Probe in ICU Patients. A Randomized Controlled Trial
Brief Title: C-MAC Videolaryngoscope for Insertion of a Transesophageal Echocardiography Probe in ICU Patients
Acronym: VIDLARECO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, Clinical Professor, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CEIG 2020/375
Record Dates: First submitted 2021-07-21; First posted 2021-07-28 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Critical Illness
Keywords: transesophageal; echocardiography; videolaryngoscope;
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: After TEE insertion, the pharyngeal mucosa will be evaluated with de C-MAC videolaryngoscope by an anesthesiologist who were blinded to the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional blind insertion technique. (Active Comparator): Transesophageal echocardiography probe will be inserted using a conventional blind insertion technique.
  Interventions: Device: Blind insertion technique
- C-MAC videolaryngoscope insertion technique (Experimental): Transesophageal echocardiography probe will be inserted using a C-MAC videolaryngoscope insertion technique to advance into esophagus under direct vision.
  Interventions: Device: C-MAC videolaryngoscope insertion technique

INTERVENTIONS:
Device: Blind insertion technique — Transesophageal echocardiography probe will be inserted using a conventional blind insertion technique.
  Arms: Conventional blind insertion technique.
Device: C-MAC videolaryngoscope insertion technique — Transesophageal echocardiography probe will be inserted using a C-MAC videolaryngoscope insertion technique
  Arms: C-MAC videolaryngoscope insertion technique

SUMMARY:
Transesophageal echocardiography (TEE) is commonly used in operating room (cardiac surgery), as well as in other critical care settings. A recent meta-analysis including only three randomized studies demonstrated that the use of a videolaryngoscope for transesophageal echocardiography probe insertion in anesthetized patients undergoing open cardiac surgery was associated with a significant reduction in the number of attempts. insertion and complications rate, compared with blind insertion or a laryngoscope-assisted insertion.

ICU patients are usually intubated, with multiple complications, requiring high doses of catecholamines, and with frequent coagulation disorders. Many of these patients, during their stay in the ICU, require a transesophageal echocardiogram. On multiple occasions, due to the critical situation of the patients, due to edema, and coagulation alteration, the placement of the echocardiography probe can be difficult, leading to complications, such as gastric bleeding or lesions in the oropharyngeal mucosa.

To avoid complications during the insertion of the TEE tube, the investigators consider it necessary to introduce it in the fewest possible attempts.

The primary aim of the present study was to compare the success rate of TEE probe insertion at the first attempt betweenn the C-MAC videolaryngoscope assisted insertion and the blind insertion technique.

The secondary aim was to compared differences between the 2 groups in the incidence of complications ( oropharyngeal mucosal injury, hematoma, ….), overall success rate, the number of insertion attempts, and the duration of insertions.

DETAILED DESCRIPTION:
One hundred intubated ICU adult patients that require transesophageal echocardiography insertion, will be randomized by means of a computer-generated randomization order into two groups: Conventional group (Group Blind), and videolaryngoscope group (group C-MAC).

Success rate of the selected technique (first attempt), overall success rate, number of attempts, complications, and duration of insertion for technique will be noted.

ELIGIBILITY:
Inclusion Criteria:

* ICU intubated patients that require transesophageal echocardiography probe insertion

Exclusion Criteria:

* patients younger than 18 years and older than 85 years
* oropharengeal infection
* esophageal injury and anatomic abnormalities
* Consent refusal for participating in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Difference in the first attempt success rate (percentage) | Participants will be followed from the beginning of the transesophageal echocardiography probe insertion through the mouth to the confirmation of successful insertion (10 minutes or three attempts)
  To compare the difference in the first attempt (percentage) of different techniques for insertion of transesophageal echocardiography probe.

SECONDARY OUTCOMES:
Difference in the overall success rate (percentage) | Participants will be followed from the beginning of the transesophageal echocardiography probe insertion through the mouth to the confirmation of successful insertion (10 minutes or three attempts)
  To compare the difference overall success rate (percentage) of different techniques for insertion of transesophageal echocardiography probe.
Difference in the incidence of complications (percentage) | Participants will be followed from the beginning of the transesophageal echocardiography probe insertion through the mouth to the confirmation of successful insertion (10 minutes or three attempts) and in the next 24 hours.
  To compare the difference in complications of different techniques for insertion of transesophageal echocardiography probe.
Difference in the duration of insertion | Participants will be followed from the beginning of the transesophageal echocardiography probe insertion through the mouth to the confirmation of successful insertion (10 minutes or three attempts) and in the next 24 hour and in the next 24 hours.
  To compare the duration of different techniques for insertion of intransesophageal echocardiography probe.

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada, Principal Investigator — University Clinical Hospital of Santiago de Compostela
Locations (1):
- Manuel Taboada, Santiago de Compostela, La Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data types: Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved T ypes of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Ishida T, Kiuchi C, Sekiguchi T, Tsujimoto T, Kawamata M. McGRATH MAC video laryngoscope for insertion of a transoesophageal echocardiography probe: A randomised controlled trial. Eur J Anaesthesiol. 2016 Apr;33(4):263-8. doi: 10.1097/EJA.0000000000000367. PMID 26575010
- [Background] Kavrut Ozturk N, Kavakli AS. Use of McGrath MAC Videolaryngoscope to Assist Transesophageal Echocardiography Probe Insertion in Intubated Patients. J Cardiothorac Vasc Anesth. 2017 Feb;31(1):191-196. doi: 10.1053/j.jvca.2016.03.150. Epub 2016 Mar 31. PMID 27498268
- [Background] Kumamoto T, Tashima K, Hiraoka C, Ikuta Y, Yamamoto T. McGRATH MAC video laryngoscope assistance during transesophageal echocardiography may reduce the risk of complications: a manikin study. BMC Anesthesiol. 2021 Jan 11;21(1):14. doi: 10.1186/s12871-020-01231-3. PMID 33430768
- [Background] Kim MK, Park SW, Sim Y, Lee JW. Use of a McGrath Videolaryngoscope to assist transesophageal echocardiography probe insertion in anesthetized patients. J Cardiothorac Vasc Anesth. 2015 Apr;29(2):e16-7. doi: 10.1053/j.jvca.2014.09.007. Epub 2014 Dec 24. No abstract available. PMID 25543216
- [Derived] Taboada M, Carinena A, Estany-Gestal A, Iglesias-Alvarez D, Veiras S, Martinez A, Eiras M, De Miguel M, Selas S, Martinez-Monzonis A, Pereira P, Bastos-Fernandez M, Gonzalez-Salvado V, Alvarez-Barrado M, Ferreiroa E, Caruezo V, Costa J, Naveira A, Otero P, Adrio B, Martinez-Cereijo JM, Fernandez A, Gonzalez-Juanatey JR, Alvarez J, Seoane-Pillado T. Videolaryngoscope versus conventional technique for insertion of a transesophageal echocardiography probe in intubated ICU patients (VIDLARECO trial): A randomized clinical trial. Anaesth Crit Care Pain Med. 2024 Apr;43(2):101346. doi: 10.1016/j.accpm.2024.101346. Epub 2024 Jan 24. PMID 38278357